CLINICAL TRIAL: NCT06837207
Title: Safety and Efficacy Study of Precise Transcranial Magnetic Stimulation for Depression Based on Individualized Functional Connectivity Localization of Orbital Frontal Cortex-habenula
Brief Title: Precision Transcranial Magnetic Stimulation for Depression Based on Orbital Frontal Cortex-habenula Circuitry
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20242429
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Depression; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individualized transcranial magnetic stimulation (Experimental)
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Individualized transcranial magnetic stimulation of targets based on the association between the orbitofrontal cortex and the functional activity of the habenula .

SUMMARY:
Thirty depressed patients will be recruited to select individualized transcranial magnetic stimulation targets based on individual orbital frontal cortex and habenula functional activity connectivity for 10 or 20 treatments to assess the efficacy and safety of this intervention

ELIGIBILITY:
Inclusion Criteria:

* Gender is not limited, age 18～60 years old;
* Comply with the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5) of the United States of America;
* Hamilton rating scale for depression (HAMD) 17-item score ≥ 18;
* The medication/psychotherapy received by the subject prior to the start of the study remained stable for at least 4 weeks .

Exclusion Criteria:

* History of serious somatic diseases or diseases that may affect the central nervous system (e.g., tumors, syphilis, etc.);
* Neurological disorders or risk of seizures, such as previous craniosynostosis, head trauma, alcoholism, abnormal electroencephalograms, MRI evidence of structural abnormalities in the brain, or family history of epilepsy;
* Patients with bipolar disorder and depression due to other psychiatric disorders (e.g., psychoactive and non-dependent substances);
* Contraindications to MRI scanning or transcranial magnetic stimulation therapy, such as metal or electronic devices placed in the body (intracranial metal foreign bodies, cochlear implants, pacemakers and stents and other metal foreign bodies), space phobia;
* People with psychotic symptoms requiring joint application of antipsychotic drugs;
* Those with high risk of suicide, or those who have already committed suicide or serious self-injury behavior requiring urgent intervention;
* Those who are pregnant, breastfeeding or planning to become pregnant during the trial;
* Other conditions judged by the investigator to be unsuitable as research subjects.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to treatment day 10 | Baseline and treatment day 10
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a widely used clinical assessment tool designed to measure the severity of depressive symptoms.The MADRS consists of 10 items, each of which addresses a different aspect of depression, such as low mood, loss of interest, sleep disorders, appetite, concentration, fatigue, inability to feel pleasure, pessimistic thinking, and suicidal ideation. Each item is scored according to the severity of symptoms, ranging from 0 to 6, with a total score ranging from 0-60, with higher scores indicating more severe depressive symptoms.
  Change = (treatment day 10 Score -Baseline Score).

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a widely used clinical assessment tool designed to measure the severity of depressive symptoms.The MADRS consists of 10 items, each of which addresses a different aspect of depression, such as low mood, loss of interest, sleep disorders, appetite, concentration, fatigue, inability to feel pleasure, pessimistic thinking, and suicidal ideation. Each item is scored according to the severity of symptoms, ranging from 0 to 6, with a total score ranging from 0-60, with higher scores indicating more severe depressive symptoms.
  Change = (28 days after the end of treatment Score -Baseline Score).
Change in Hamilton Anxiety Scale scores from baseline to treatment day 10 | Baseline and treatment day 10
  Hamilton Anxiety Scale (HAMA）is suitable for assessing the severity of anxiety symptoms. It has 14 items and adopts a 5-level scoring method of 0-4 points.Possible scores range from 0 to 56 and the higher the score, the worse the symptom.
  Change = (treatment day 10 Score -Baseline Score).
Change in Hamilton Anxiety Scale scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  Hamilton Anxiety Scale (HAMA）is suitable for assessing the severity of anxiety symptoms. It has 14 items and adopts a 5-level scoring method of 0-4 points.Possible scores range from 0 to 56 and the higher the score, the worse the symptom.
  Change = (28 days after the end of treatment Score -Baseline Score).
Change in Hamilton Depression Scale（HAMD-17）scores from baseline to treatment day 10 | Baseline and treatment day 10
  Hamilton Depression Scale（HAMD-17） is a commonly used clinical evaluation standard for the severity of depressive symptoms. There are 17 items in total, which can be scored before and after treatment to evaluate the severity of the disease and the treatment effect.Possible scores range from 0 to 52 and the higher the score, the worse the symptom.
  Change = (treatment day 10 Score -Baseline Score).
Change in Hamilton Depression Scale（HAMD-17）scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  Hamilton Depression Scale（HAMD-17） is a commonly used clinical evaluation standard for the severity of depressive symptoms. There are 17 items in total, which can be scored before and after treatment to evaluate the severity of the disease and the treatment effect.Possible scores range from 0 to 52 and the higher the score, the worse the symptom.
  Change = (28 days after the end of treatment Score -Baseline Score).
Change in Pittsburgh sleep quality index (PSQI) scores from baseline to treatment day 10 | Baseline and treatment day 10
  The Pittsburgh Sleep Quality Index is suitable for patients with sleep disorders to evaluate the quality of their sleep, as well as for the general population to assess the quality of their sleep. The scale consists of 9 questions, of which the first 4 are fill-in-the-blanks and the last 5 are multiple-choice (question 5 contains 10 sub-questions) Change = (treatment day 10 Score -Baseline Score).
Change in Pittsburgh sleep quality index (PSQI) scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  The Pittsburgh Sleep Quality Index is suitable for patients with sleep disorders to evaluate the quality of their sleep, as well as for the general population to assess the quality of their sleep. The scale consists of 9 questions, of which the first 4 are fill-in-the-blanks and the last 5 are multiple-choice (question 5 contains 10 sub-questions) Change = (28 days after the end of treatment Score -Baseline Score).
Change in Snaith-Hamilton Pleasure Scale scores from baseline to treatment day 10 | Baseline and treatment day 10
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a self-report questionnaire used to assess pleasure deficits (anhedonia).The SHAPS scale consists of 14 entries asking subjects to rate their level of agreement with pleasure responses in a number of pleasurable situations on a 4-point scale. The measure taken is the subject's situation in the most recent period of time. Pleasure experience is measured in four domains: interests/recreation, social interactions, sensory experiences, and food/drink. The scale has good reliability and validity in normal as well as clinical populations. Each entry is rated on a 4-point scale, with "strongly agree, agree, disagree, and strongly disagree" scoring from 1 to 4, respectively.
  Change = (treatment day 10 Score -Baseline Score).
Change in Snaith-Hamilton Pleasure Scale scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a self-report questionnaire used to assess pleasure deficits (anhedonia).The SHAPS scale consists of 14 entries asking subjects to rate their level of agreement with pleasure responses in a number of pleasurable situations on a 4-point scale. The measure taken is the subject's situation in the most recent period of time. Pleasure experience is measured in four domains: interests/recreation, social interactions, sensory experiences, and food/drink. The scale has good reliability and validity in normal as well as clinical populations. Each entry is rated on a 4-point scale, with "strongly agree, agree, disagree, and strongly disagree" scoring from 1 to 4, respectively.
  Change = (28 days after the end of treatment Score -Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: Huaning Wang, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139
- [Background] Philip NS, Barredo J, van 't Wout-Frank M, Tyrka AR, Price LH, Carpenter LL. Network Mechanisms of Clinical Response to Transcranial Magnetic Stimulation in Posttraumatic Stress Disorder and Major Depressive Disorder. Biol Psychiatry. 2018 Feb 1;83(3):263-272. doi: 10.1016/j.biopsych.2017.07.021. Epub 2017 Aug 8. PMID 28886760
- [Background] Cash RFH, Weigand A, Zalesky A, Siddiqi SH, Downar J, Fitzgerald PB, Fox MD. Using Brain Imaging to Improve Spatial Targeting of Transcranial Magnetic Stimulation for Depression. Biol Psychiatry. 2021 Nov 15;90(10):689-700. doi: 10.1016/j.biopsych.2020.05.033. Epub 2020 Jun 7. PMID 32800379
- [Background] Goldstein-Piekarski AN, Ball TM, Samara Z, Staveland BR, Keller AS, Fleming SL, Grisanzio KA, Holt-Gosselin B, Stetz P, Ma J, Williams LM. Mapping Neural Circuit Biotypes to Symptoms and Behavioral Dimensions of Depression and Anxiety. Biol Psychiatry. 2022 Mar 15;91(6):561-571. doi: 10.1016/j.biopsych.2021.06.024. Epub 2021 Jul 11. PMID 34482948